CLINICAL TRIAL: NCT01108107
Title: Neoadjuvant Chemotherapy and Biological Treatment for Patients With Locally Advanced Colon Cancer
Brief Title: Neoadjuvant Treatment of Colon Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: S-20100014
Record Dates: First submitted 2010-04-14; First posted 2010-04-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2014-03

CONDITIONS: Colon Cancer
Keywords: Colon cancer; Neoadjuvant treatment; KRAS mutation; BRAF mutation; PIK3CA mutation; Possibly avoid chemotherapy after operation
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin; Capecitabine; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy only (Other): Chemotherapy only, if mutations in KRAS, BRAF or PIK3CA gene
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine
- Chemotherapy + biological treatment (Other): Addition of biological treatment, if no mutations in KRAS, BRAF, and PIK3CA genes.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Biological: Panitumumab

INTERVENTIONS:
Drug: Oxaliplatin — 130 mg/m2 intravenously on day 1 of a 3-weekly cycle
  Arms: Chemotherapy only
Drug: Capecitabine — 2000 mg/m2/day (tablets) on day 1 and 14 of a 3-weekly cycle
  Arms: Chemotherapy only
Drug: Oxaliplatin — 130 mg/m2 intravenously on day 1 of a 3-weekly cycle
  Arms: Chemotherapy + biological treatment
Drug: Capecitabine — 2000 mg/m2/day (tablets) on day 1 and 14 of a 3-weekly cycle
  Arms: Chemotherapy + biological treatment
Biological: Panitumumab — 9 mg/kg intravenously on day 1 of a 3-weekly cycle
  Arms: Chemotherapy + biological treatment

SUMMARY:
This study will investigate

* the effect of preoperative combination chemotherapy in patients with locally advanced colon cancer with mutation in the KRAS, BRAF or PIK3CA gene
* the effect of preoperative combination chemotherapy in combination with biological treatment in patients without mutation in the KRAS, BRAF or PIK3CA gene.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified locally advanced T3 or T4 colon cancer assessed by CT scan
* Analysis of KRAS, BRAF, PIK3CA
* Age ≥18 år
* Performance status ≤ 2
* Hematology

  * ANC ≥ 1.5x10^9/l. Thrombocytes ≥ 100x10^9/l.
* Biochemistry

  * Bilirubinaemia ≤ 3 x UNL. ALAT ≤ 5 x UNL
* Consent to translational research
* Fertile women must present a negative pregnancy test and use secure birth control during and 3 months after treatment.
* Written and orally informed consent.

Exclusion Criteria:

* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment, active severe infections or other concurrent disease.
* Peripheral neuropathy NCI grade >1
* Other malignant disease within 5 years prior to enrollment, except basal cell squamous carcinoma of the skin and cervical carcinoma-in-situ
* Other investigational treatment within 30 days prior to treatment start
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* Bleeding tumors
* Hypersensitivity to one or more of the substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The frequency of patients requiring adjuvant chemotherapy based on the histological evaluation of the preparation from the operation. | Within 1 week after surgery

SECONDARY OUTCOMES:
Recurrence free survival | Up to 2 years.
Overall survival | Up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, DMSc, Principal Investigator — Vejle Hospital
Locations (3):
- Denmark (3):
  - Department of Oncology, Herlev Hospital, Herlev
  - Dept. of Oncology, Hilleroed Hospital, Hilleroed
  - Department of Oncology, Vejle Hospital, Vejle

REFERENCES:
- [Derived] Dam C, Lund-Rasmussen V, Ploen J, Jakobsen A, Rafaelsen SR. Computed tomography assessment of early response to neoadjuvant therapy in colon cancer. Dan Med J. 2015 Jul;62(7):A5103. PMID 26183044